CLINICAL TRIAL: NCT02721225
Title: Promoting Healthy Foetal and Post Natal Growth by Modulating Vaginal or Gut Micro Biota With Supplementation of Prebiotic Agent ( Fructooligosaccharide) in Pregnant Women- a Randomized Double Blind Community Based Clinical Trial.
Brief Title: Prebiotic in Preventing Low Birth Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Karolinska Institutet (Other); Swedish International Development Cooperation Agency (SIDA) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PR-14038
Record Dates: First submitted 2016-03-14; First posted 2016-03-29 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2018-08

CONDITIONS: Birth Weight <2500gm; Genitourinary Tract Infection
MeSH Terms: interventions — fructooligosaccharide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fructooligosaccharide (Active Comparator): One kind of prebiotics agent defined as "selectively fermented ingredients that allow specific changes, both in the composition and/or activity in the gastrointestinal microbiota that confers benefits upon host well-being and health"
  Interventions: Dietary Supplement: Fructooligosaccharide
- Pocari-Sweat (Placebo Comparator): Commercially produced isotonic solution by Otsuka Pharmaceutical Co., Ltd., Tokyo,Japan
  Interventions: Dietary Supplement: Pocari-Sweat

INTERVENTIONS:
Dietary Supplement: Fructooligosaccharide — A prebiotics defined as "selectively fermented ingredients that allow specific changes, both in the composition and/or activity in the gastrointestinal microbiota that confers benefits upon host well-being and health"
  Arms: Fructooligosaccharide
Dietary Supplement: Pocari-Sweat — Commercially used isotonic solution produced by Otsuka Pharmaceuticals Co. Ltd., Tokyo, Japan.
  Arms: Pocari-Sweat

SUMMARY:
More than 20 million infants worldwide, representing 16 per cent of all births, are born with low birth weight, 96 per cent of them in developing countries. Bangladesh having one of the highest incidence rate (21.6%) in the world.The short-term consequences of LBW is 12 times higher perinatal mortality. It is estimated that LBW causes 60 to 80 % of neonatal deaths. For the survivors, the effects are long lasting and largely irreversible. Infants born LBW are at 2-4 times greater risk to develop acute diarrhea, pneumonia or acute respiratory tract infection than their normal birth weight counterparts. Adults born with LBW suffer increased risk of high blood pressure, coronary heart disease (CHD), non insulin dependent diabetes mellitus, obstructive lung diseases, or renal damage.

Genitourinary (GU) infection, as a major risk factor for low birth weight deliveries affecting a very large number of women both in the industrialized and the developing world. In Bangladesh, there was a high incidence of UTI in 21-25 years age group (44.61%). The bottom line for GU infection is that lactobacilli, healthy bacteria lose their dominant. Recently, the protective role of the commensal microbiota has come into focus for its infection-inhibiting function. Lactobacilli that colonize the gastrointestinal tract or vagina can either significantly modulate the colonic microbiota by increasing the number of specific prebiotic bacteria such as lactobacilli and bifidobacteria or reducing undesired intestinal colonization of pathogenic bacteria. Prebiotic like Fructooligosaccharide (FOS) is known to promote growth of normal healthy flora like lactobacilli (LAB). FOS supplementation in early pregnancy improves vaginal or gut microflora with LAB , which will control GU infection and improve pregnancy outcome and promote infant's growth and development

DETAILED DESCRIPTION:
Medical research over the last ten years has identified genitourinary (GU) infection, as a major risk factor for low birth weight deliveries affecting a very large number of women both in the industrialized and the developing world. It is estimated that up to about 1 billion of women are affected annually by urinary infections worldwide. Urinary tract infections (UTI) are also most common bacterial infections during pregnancy. In Bangladesh, there was a high incidence of UTI in 21-25 years age group (44.61%). The bottom line for GU infection is that lactobacilli, healthy bacteria lose their dominant.

The role of normal vaginal micro-biota in urogenital health Recently, the protective role of the commensal microbiota has come into focus for its infection-inhibiting function. Lactobacilli are now the favourite probiotic ("health promoting") bacteria. There are clinical evidence to show that Lactobacillus strains GR-1 and RC-14 were shown to reduce UTI, BV and infections associated with yeast pathogens.

Fructoligosacharride, a prebiotic agent At present, considerable attention is focused on determining ways to increase the number of probiotic microorganisms including lactobacilli that colonize the gastrointestinal tract or vagina. Prebiotics are substances that can either significantly modulate the colonic microbiota by increasing the number of specific probiotic bacteria such as lactobacilli and bifidobacteria or reducing undesired intestinal colonization of pathogenic bacteria by mimicking their attachment sites on the intestinal mucosa.

Design and methods In a, double- blind, placebo- controlled study, 210 early pregnant community women (6-12 weeks gestation) will be randomized to either FOS or placebo, administered orally, 6g/day for 6 months. Vaginal smear and urine samples will be followed for LAB using Nugent's score and to exclude UTI respectively. Birth events including weight will be documented. Stool or nasopharyngeal samples from their infants will be obtained at week-24, 30, and 36 to see levels of LAB. Anthropometry and diseases morbidity will be monitored during infancy.

Outcome measures/variables:

* Primary: 1. Incidence of LBW (birth weight below 2500 gram)
* Secondary 1. Rate of vaginal and intestinal colonization of LAB and/or GU infection at week 12, 24, 36 gestation and gain in z-score (weight for height, weight for age and height for age) of infant from birth

ELIGIBILITY:
Inclusion Criteria:(i) Age: 18-35 years (ii) Missed period : 6-12 weeks (iii) Positive pregnancy test by dip stick method in a morning urine sample (iv) Parity: any but with history of previous normal delivery (v) Weight: Body Mass Index greater than 18.5 but less than 35 (vi) Past obstetric history: Uncomplicated pregnancy, unremarkable medical and obstetric Conditions. (vii) Written informed consent witnessed by husband or legal guardian (thumb impression for those who are illiterate)

Exclusion Criteria:

Exclusion criteria The exclusion criteria will be (i) known previous H/O gestational diabetes and pre-eclamptic toxaemia (PET), (ii) any systemic disorder or chronic illness (iii) history of previous major gynaecological problem or treatment i.e., myomectomy, hysterotomy, knife cone biopsy etc.

(iv) uterine/vaginal abnormality or (v) 3 or more previous consecutive spontaneous abortions and no subsequent non vaginal delivery, etc.).

(vi) Hb level ( < 7 gm/dL), and/or oedema (vii) History of taking antibiotic within 3 weeks prior to this study (viii) Complications in previous pregnancy (stillbirth, preterm labour, complicated instrumental delivery, retained placenta, 3°/ 4° perineal tear, transverse lie, placental abruption, Previous baby of <2.5 kg / >4.5 kg) (ix) Women unwilling to comply with study protocol (x) Presence of UTI or bacteriuria in a morning mid stream fresh urine sample (xi) Presence of abnormal vaginal flora (Nugent score >7) (xii) History of irregular bleeding due to injectable Depo-Provera

-

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
1. Infant birth weight | just after birth
  Normal Birth Weight is equal or more than 2500 gm and low birth weight is less than 2500gm
Gestational age | upto 40 weeks of pregnancy
  Gestational age measured in weeks from the first day of women's Last menstrual period to the current date.
  Delivery before 36 weeks of pregnancy will be considered as premature

SECONDARY OUTCOMES:
Vaginal colonization of Lactobacillus (LAB) | at 12, 18 and 30 weeks of gestation
  Collection of vaginal swab to see colonization of LAB and also Nugent score Nugent score less than 7 indicate normal condition and equal or more than 7 indicates Bacterio-vaginal infection
Intestinal Colonization of LAB | at 12, 24 and 36 weeks of gestation from pregnant women and at birth from the infant
  Collection of stool to see colonization of LAB
Rate of Genito-urinary (GU) infection | at 12, 18, 24 and 36 weeks of pregnancy
  Collection of urine for culture to see any infection. If bacterial colony count >10to the power 5 indicates genito urinary infection
Gain in Z-score of infant from birth | from birth to 3 months of age of infant
  According to WHO weight for length and weight for age (50th percentile) reference table
Incidence of Acute respiratory infection and diarrhoea | From birth to 3 months of age
  Fever, cough, respiratory distress,chest indrawing etc and passsage of loose stool

CONTACTS AND LOCATIONS:
Overall Officials: Shafiqul A Sarker, MD, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Shafiqul Alam Sarker, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided